CLINICAL TRIAL: NCT04740008
Title: Impact of Low Nicotine Cigarette Messaging on Risk Perceptions and Hypothetical Tobacco and Nicotine Product Choices.
Brief Title: Impact of Low Nicotine Cigarette Messaging on Perceptions and Cigarette Choices
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPH-2020-29384; 2020LS214 (Other: University of Minnesota Masonic Cancer Center)
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Smoking; Cigarette
Keywords: Low Nicotine Content; Educational Messaging; Cigarette; Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control message on low nicotine cigarettes (Experimental)
  Interventions: Drug: Low Nicotine Content Cigarettes; Other: Control message
- Test message on low nicotine cigarettes (Experimental)
  Interventions: Drug: Low Nicotine Content Cigarettes; Other: Test message

INTERVENTIONS:
Drug: Low Nicotine Content Cigarettes — Low Nicotine Content Cigarettes 0.4 mg/g nicotine; 9 mg tar Other Name: Reduced Nicotine Content Cigarettes
Other: Control message — Participants will read control message
  Arms: Control message on low nicotine cigarettes
Other: Test message — Participants will read test message
  Arms: Test message on low nicotine cigarettes

SUMMARY:
The purpose of this research is to evaluate the effects of low nicotine content cigarette (LNC) educational messaging on perceptions of low nicotine cigarettes, tobacco/nicotine product choice preferences (hypothetical), LNC cigarette subjective ratings, and LNC cigarette abuse liability among adult smokers.

DETAILED DESCRIPTION:
This randomized single-site study will assess the subject's risk perceptions and hypothetical tobacco product choices based on their exposure to an educational messaging condition related to nicotine content in cigarettes.

Subjects (N=40 in each group) will be given a pack of low nicotine content cigarettes (LNC; 0.4 mg/g) and will be randomly assigned to read one of two messaging conditions on low nicotine cigarettes.

Smokers will undergo a telephone screening to assess eligibility, then move on to the next steps of the study depending on eligibility:

1. Virtual Zoom Screening - Completed after telephone screen: Informed consent is obtained and then an interview where data is collected and eligibility is further assessed.
2. Curbside Visit - Completed after the screening and if eligible: Breath test, and if necessary a urine test, is performed to assess smoking levels and urine pregnancy test is attained (if applicable). If eligible, randomization to messaging condition occurs and participants provided a pack of low nicotine content cigarettes.
3. Virtual Zoom Home Session - Completed after curbside and if eligible based on curbside: Surveys assessing main outcome variables assessed.
4. Follow-up - Completed 1 week after the virtual Zoom session: Interview where assessment of health and product usage is assessed.

Except for the initial telephone screening, participants will receive compensation for each part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* At least 21 years of age
* Biochemically confirmed smoker

Exclusion Criteria:

* Unstable health condition
* Unstable medications
* Pregnant or nursing
* Unreliable access to a computer, smart phone or tablet without working camera and internet access for telehealth visits and online questionnaires

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
Proportion of participants that choose ANDS or no tobacco | Within 17 days of virtual screening
  Proportion of participants who select to use ANDS or no tobacco if LNC cigarettes were the only cigarettes available will be compared in arm 1 versus arm 2

CONTACTS AND LOCATIONS:
Overall Officials: Dana Mowls Carroll, Ph.D., M.P.H, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota, Tobacco Research Program, 717 Delaware St., SE, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Intend to share findings from this research through publications and presentations. Institutions and individuals wishing to access any resources or data must contact the Principal Investigator (Carroll). Data will be available in two formats. One will be a summary of the data, with graphs and tables, posted as pdf files and as raw individual-level data for analysis. Data generated by this grant will be made to outside investigators, according to NIH Guidance. When data are shared, there will be no limits placed on how the data will be used. Users will agree, however, that the recipient must not transfer the data to other users and that the data are only to be used for research purposes. A record of transfer of data and a copy of the dataset that was distributed will be kept by University of Minnesota
Time Frame: Data will not be available until primary and secondary papers are accepted for publication.
Access Criteria: Persons requesting data must do so in writing, identifying their affiliation and how the data will be used. Upon review, access will be determined.